CLINICAL TRIAL: NCT02566343
Title: Preoperative Diagnostic Tests for Pulmonary Risk Assessment in Patients With Chronic Obstructive Pulmonary Disease (COPD) Undergoing Major Surgery
Brief Title: Preoperative Diagnostic Tests for Pulmonary Risk Assessment in COPD
Acronym: PredicT
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV4743
Record Dates: First submitted 2015-09-21; First posted 2015-10-02 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2016-06

CONDITIONS: Lung Diseases, Obstructive; Postoperative Complications
Keywords: Spirometry; Exercise Test; Blood Gas Analysis; Respiratory Function Tests; Diagnostic Techniques, Respiratory System; Surgical Procedures, Operative
MeSH Terms: conditions — Lung Diseases, Obstructive; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD cohort: confirmed COPD: 240 patients with COPD confirmed by spirometry undergoing high-risk noncardiac major surgery in the University Medical Center Hamburg-Eppendorf will be included in this group.
- Control cohort: disproved COPD: 80 patients without COPD (clinical risk factors but negative spirometry) undergoing high-risk noncardiac major surgery will be included as a control group.

SUMMARY:
This prospective study intends to investigate the incidence of postoperative pulmonary complications (PPC) or in-hospital mortality in patients with COPD or at risk for COPD undergoing high-risk noncardiac major surgery and to identify relevant risk factors. This study aims to quantify and compare the diagnostic performance of preoperative functional tests, exercise capacity, clinical assessment tests and predictive scoring systems to predict PPC or in-hospital mortality in these patients.

DETAILED DESCRIPTION:
COPD is associated with high perioperative morbidity and mortality and PPC frequently occur in these patients. However, concepts for preoperative pulmonary risk assessment and the predictive value of routine preoperative exercise capacity, clinical assessment and pulmonary function tests are still poorly characterized.

Objectives:

* To determine the incidence of the composite end point of PPC or all cause in-hospital mortality in patients with confirmed COPD (spirometry) and patients with clinical risk factors in whom spirometry disproved COPD.
* To determine the predictive value of exercise capacity, clinical assessment tests, pulmonary function tests and predictive scoring systems to predict the composite end point in these patients.
* To identify relevant risk factors and predictors associated with the composite end point.

Methodology:

Prospective single-centre observational study

All patients receive a structured preoperative pulmonary risk assessment with:

1. standardized clinical questionnaire
2. COPD Assessment Test (CAT™)
3. exercise capacity (symptom-limited stair climbing)
4. spirometry
5. capillary blood gas Analysis

Postoperative follow-up is planned between the 2nd and 5th day after extubation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* High-risk noncardiac major surgery with an anticipated operation time ≥ 120 minutes and/or planned postoperative intensive care unit admission
* Typical clinical signs for COPD (dyspnea, chronic cough, chronic sputum production, exposure to risk factors)
* Confirmed COPD (medical history) or clinical risk factors for COPD
* Positive COPD Assessment Test (CAT™)

Exclusion Criteria:

* < 18 Years
* Pregnancy
* Lack of cooperation
* Inability to provide functional tests like spirometry or stairclimbing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for major surgery, who present in the pre-assessment clinic of the University Medical Center Hamburg-Eppendorf during the study recruitment period, will be screened for eligibility. Patients with typical clinical signs and a positive COPD Assessment Test (CAT™) qualify for spirometry. After informed consent 80 patients with disproved COPD (FEV1/FVC ratio ≥ 0.70) and 240 patients with confirmed COPD (FEV1/FVC ratio < 0.70) will consecutively be analysed.
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Composite end point of postoperative pulmonary complications (PPC) or all cause in-hospital mortality | until hospital discharge up to 6 months after surgery

SECONDARY OUTCOMES:
Forced expiratory volume in one second to forced vital capacity ratio (FEV1/FVC) and FEV1 % predicted | within 1 week after extubation
Carbon dioxide (pCO2) and oxygen (pO2) partial pressures from blood gas analysis | within 1 week after extubation
Postoperative new respiratory symptoms (e.g. dyspnea or wheezing) or treatment for exacerbation (e.g. new systemic glucocorticosteroids or bronchodilators) | until hospital discharge up to 6 months after surgery
New pulmonary radiological findings (e.g. pneumonia or pneumothorax) | until hospital discharge up to 6 months after surgery
Duration of hospitalization (days) | until hospital discharge up to 6 months after surgery
Duration of postoperative respirator support (h) | until hospital discharge up to 6 months after surgery
Length of stay in the intensive care unit (days) | until hospital discharge up to 6 months after surgery
Frequency of unplanned intensive care unit admission, prolonged oxygen requirement, reintubation, non-invasive ventilation (NIV) or extracorporeal lung assist | until hospital discharge up to 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Christian Zöllner, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta H, Ramanan B, Gupta PK, Fang X, Polich A, Modrykamien A, Schuller D, Morrow LE. Impact of COPD on postoperative outcomes: results from a national database. Chest. 2013 Jun;143(6):1599-1606. doi: 10.1378/chest.12-1499. PMID 23287892